CLINICAL TRIAL: NCT03874767
Title: Can Mobility Technicians Provide Value to Hospitalized Patients?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Bandwidth and logistics issues exacerbated by COVID-19 pandemic
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Heather Skaar, Administrative Director, Physical Medicine & Rehabilitation Acute Care, Dayani Center, Orthopaedic Therapy, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 000000000
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Hip Fractures; Lower Extremity Fracture; Lung Transplant
Keywords: patient mobility; ambulation
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: single center, pragmatic cluster trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10th floor south (Active Comparator): The unit in this arm will be assigned physical therapists plus mobility technicians in the first month and only physical therapists in the following month.
  During months where a unit has been assigned the mobility technicians, the mobility technician, along with nursing staff, will deliver additional prescribed mobility as well as standard-of-care prescribed therapy provided by physical therapy staff:
  1. On evaluation, a PT will assign a JH-HLM scale rating to the patient
  2. If the score is 4 or higher, the PT will add the patient to the mobility technician patient list
  3. The mobility technician will then see that patient daily, unless the score is <4
  4. Each PT session will involve a re-assessment by the PT of the JH-HLM scale rating as well as the Function Independence Measurement (FIM) score, and subsequently will update the recommended therapy if appropriate
  5. The mobility technician will work with PT and nursing to determine the best time to deliver mobility
  Interventions: Behavioral: Patient Mobility
- 6th floor Round Wing (Active Comparator): The unit in this arm will be assigned only physical therapists in the first month and physical therapists plus mobility technicians in the following month.
  During months where a unit has been assigned the mobility technicians, the mobility technician, along with nursing staff, will deliver additional prescribed mobility as well as standard-of-care prescribed therapy provided by physical therapy staff:
  1. On evaluation, a PT will assign a JH-HLM scale rating to the patient
  2. If the score is 4 or higher, the PT will add the patient to the mobility technician patient list
  3. The mobility technician will then see that patient daily, unless the score is <4
  4. Each PT session will involve a re-assessment by the PT of the JH-HLM scale rating as well as the Function Independence Measurement (FIM) score, and subsequently will update the recommended therapy if appropriate
  5. The mobility technician will work with PT and nursing to determine the best time to deliver mobility
  Interventions: Behavioral: Patient Mobility

INTERVENTIONS:
Behavioral: Patient Mobility — A team of two mobility technicians will switch between two units on a monthly basis. The unit staffed by the mobility technician will be referred to as the intervention unit, while the other will be referred to as the control unit. One unit will start as the control unit and will switch to being the intervention unit after one month. Similarly, the other unit will start as the intervention unit and will switch to becoming the control unit after one month. All patients present on a unit during the intervention period will be provided mobility technician support according to standardized clinical guidelines that have been developed by the care team and described below. Patients who are present on a unit at the time of cross-over will not be included in the analysis, but will either no longer receive mobility technician support (if crossing from intervention to control) or will start to receive mobility technician support (if switching from control to intervention).

SUMMARY:
The specific aim of this study is to determine the impact of the addition of a dedicated mobility technician to the care team on specialty specific outcomes for patients recovering from surgical treatment for a hip or lower extremity long bone fracture or a lung transplant.

The practice of post-operative early ambulation has been shown to improve outcomes by promoting enhanced recovery after surgery in a variety of patients. To that end, VUMC is establishing a "Culture of Mobility". To do so, additional personnel are being hired to help ambulate patients with traumatic hip and femur fractures, other fractures of the lower extremity long bones, as well as those post-lung transplant or readmitted post-lung transplant based upon the best available evidence supporting mobility programs. The added personnel are needed as the currently available resources have insufficient bandwidth to ensure complete early ambulation for all patients. The relative effectiveness of adding a dedicated resource is assumed. Although the literature suggests adding person-hours increases the amount of mobility achieved, there is an opportunity to evaluate whether this is really the case.

The goal of this study is to evaluate the impact of adding the mobility technician to the existing care team. The mobility technician will be assisting patients who could benefit from early ambulation after surgery. We hypothesize that by adding this staffing resource, more patients will get the appropriate level of usual care. Specifically, we expect that adding the resource increases the proportion of those patients who are receiving the prescribed amount of early ambulation post-surgery, with subsequent improvements in functional independence at discharge, and decreases length of stay since patients achieve readiness for discharge sooner.

ELIGIBILITY:
Inclusion Criteria:

* All traumatic fractures of the hip or a lower extremity long bone
* Post-lung transplant patient
* Patient readmitted following a lung transplant

Exclusion Criteria:

* Non-traumatic joint replacements
* Patients with ankle fractures
* Pre-lung transplant patients
* Patients readmitted to the orthopedics unit following a traumatic injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Length of Stay | Admission to discharge (usually less than 1 week)
  The primary outcome for this study will be length of stay (LOS), defined as time from admission to the unit to discharge from the unit in days. The LOS will be obtained for this study from the Electronic Medical Record (EMR).
AM-PAC 6 Clicks score | 7 days post ICU discharge +/- 1 day for post-lung transplant patients and day 7 +/- 1 days for readmitted post-lung transplant patients. Raw scores range from 6-24, where a lower number suggests higher functional/mobile impairment.
  The AM-PAC 6 clicks score will be the co-primary outcome for this study within the transplant population and is a measurement that helps describe patient basic mobility. This score will be obtained for this study from the Electronic Medical Record (EMR)

SECONDARY OUTCOMES:
Function Independence Measurement (FIM) score | At discharge (usually less than 1 week after admission)
  Patient function is assessed using the FIM™ instrument at the start of a rehabilitation episode of care and at the end of a rehabilitation episode of care. Admission assessment is collected within 72 hours of the start of a rehabilitation episode. Discharge assessment is collected within 72 hours prior to the end of a rehabilitation episode.
  The FIM score measures a patient's mobility. The score ranges from 6 to 24, where 6 means most limited mobility and 24 means normal mobility.
Johns Hopkins Highest Level of Mobility (JH-HLM) score | At discharge (usually less than 1 week after admission)
  The JH-HLM scale was developed based on input from multiple disciplines (nursing, rehabilitation therapists, physicians, etc.) to help record the mobility that a patient actually does, standardize the description of patient mobility, and to be used as a performance measure for quality improvement projects.
  The JH-HLM score measures a patient's mobility. The score ranges from 1 to 8, where 1 means most limited mobility and 8 means normal mobility.
Total amount of mobility therapy | Admission to discharge (usually less than 1 week)
  Amount of mobility provided, which will be derived from clinical data extracted from the EMR. This will be measured through number additional mobility sessions.
Amount of ambulation | Admission to discharge (usually less than 1 week)
  Amount of ambulation achieved

CONTACTS AND LOCATIONS:
Overall Officials: Heather Skaar, PT, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD.